CLINICAL TRIAL: NCT03610633
Title: Impact of Oxytocin on Neurobiologic Substrates of Social Stress in Individuals With Alcohol Use Disorder
Brief Title: Oxytocin and Stress Response in Alcohol Use Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PRO 50913
Record Dates: First submitted 2016-02-12; First posted 2018-08-01 (Actual); Results first posted 2019-10-23 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-09

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxytocin/alcohol use disorder (Experimental): Participants will receive 24 IU of oxytocin prior to completing fMRI scanning procedures.
  Interventions: Drug: Oxytocin
- Placebo/Alcohol use disorder (Placebo Comparator): Participants will receive placebo (saline solution) prior to completing fMRI scanning procedures.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin — The neuropeptide oxytocin (OT) increases social approach, trust, and reduces anxiety to social stress.
  Other Names: Pitocin
  Arms: Oxytocin/alcohol use disorder
Drug: Placebo — Saline solution.
  Arms: Placebo/Alcohol use disorder

SUMMARY:
Individuals with alcohol use disorder (AUD) will complete one functional Magnetic Resonance Imaging (fMRI) scanning visit. Prior to the scan, individuals will receive a nasal spray of either 24 international units (IU) of oxytocin (OT), or placebo (PBO). During the scan, they will perform the Montreal Imaging Stress Task (MIST), a social stress task. Subjective craving and anxiety data will be collected.

DETAILED DESCRIPTION:
Participants: Twenty-four individuals with AUD will be recruited through the Clinical Intake and Assessment (CIA) Core of the Alcohol Research Center (ARC). Screening and basic assessments will be conducted by the CIA Core to determine eligibility and suitability for participation in this pilot project. Each individual will sign an Institutional Review Board (IRB)-approved informed consent form.

Study Visit Assessments: The Drinking Motives Questionnaire Revised will be used to assess motivation for drinking across four subscales: (1) coping motives; (2) social motives; (3) conformity motives; and (4) enhancement motives. The Form 90 will be used to assess daily alcohol consumption in the 90 days prior to the study visit and the time from last drink . A modification of the Within Session Rating Scale will be used to assess craving and mood.

Study Visit Procedures: Participants will be asked to arrive at the Addiction Sciences Division on the study visit day. Female participants will have their urine tested for pregnancy. Females who test positive for pregnancy will be excluded. All participants will be tested for drugs of abuse and alcohol. Patients testing positive for drugs, with the exception of marijuana, will be excluded; patients testing positive for alcohol may be re-scheduled. Participants will be asked about substance use in the last 90 days and will fill out the Drinking Motives Questionnaire. Subjects who have not had a research physical exam within the last 30 days will have a physical completed. They will then be escorted to the scanner at 30 Bee Street.

The study will use a double-blind placebo controlled design. Intranasal OT (n=12) or PBO (n=12) sprays will be administered at 11:30 am, approximately 45 min prior to the scanning session. This dose and timing of OT administration were selected based on the literature.

MIST Procedure: The study will use a block design of three, 6-min runs separated by 2-min of rest for feedback, for a total of 24 min. During each run, participants will be exposed to 40-sec blocks of three different conditions (rest, control, and experimental). Prior to the task, participants will are shown images of what the screen will look like during each condition. The participants will be instructed to relax during the rest condition and focus on the screen. During the control condition, the participants will be asked to answer math problems as accurately as possible but will also be told that their responses will not be recorded. During the experimental condition, the participants will be asked to perform the math task as quickly and accurately as possible. A performance bar located on the screen will allow them to see their performance as compared to an "average" person. The participants will be told that the average person would answer about 85% of the problems correctly; however, the program limits the participants' performance rate to between 35-45%. A time limit will be enforced throughout the experimental condition. After each run, the participants will be given negative feedback from the investigator.

Blood Oxygen Level Dependent (BOLD)-fMRI Procedure: Data will be acquired on a Siemens Trio 3T scanner in MUSC's Center for Biomedical Imaging. For co-registration and normalization of functional images, a high resolution T1-weighted Magnetization-Prepared Rapid Acquisition with Gradient Echo (MPRAGE) anatomical image will be acquired with the following parameters: Time of Repetition (TR)= 2100 ms, Echo Time (TE)= 4.18 ms, flip angle= 12°, field of view= 256 mm, slice thickness= 1.0 mm. The scanning planes will be oriented parallel to the anterior commissure-posterior commissure line. Participants will be asked to relax and keep their eyes opened and fixed on a cross-hair for 6 min while resting state data are collected. Participants will then complete the MIST. T2*-weighted gradient-echo planar images (EPI) will be acquired with the following parameters: TR= 2000 ms, TE= 27 ms, flip angle= 76º, matrix 64 x 64, field of view= 23 cm, slice thickness= 3.7 mm with no gap, with 36 slices to cover the entire brain.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21-40.
2. Subjects must be able to provide informed consent and function at an intellectual level sufficient to allow accurate completion of all assessment instruments.
3. Meets the DSM 5 criteria for current alcohol use disorder.
4. Reports drinking on average, at least 20 standard alcoholic drinks per week for at least the past three months.
5. Currently not engaged in, and does not want treatment for, alcohol related problems.
6. Lives within 50 miles of the study site.
7. Subjects must consent to random assignment.
8. Able to maintain abstinence for two days (without the aid of detoxification medications) as determined by self report and breathalyzer measurements Subjects must also have a negative breathalyzer urine drug screen at the study visit.
9. Subjects must consent to the study visit which includes an outpatient admission to the Addiction Sciences Division and completing one functional magnetic resonance imaging (fMRI) scanning session.

Exclusion Criteria:

1. Currently meets DSM 5 criteria for any other psychoactive substance use disorder.
2. Is determined
3. Any psychoactive substance use (except marijuana and nicotine) within the last 30 days by self-report and urine drug screen. For marijuana, no use within the last seven days by verbal report and negative (or decreasing) urine THC levels.
4. Meets DSM 5 criteria for current major depression, panic disorder, obsessive-compulsive disorder, post traumatic stress syndrome, bipolar affective disorder, schizophrenia, dissociate disorders, eating disorders, and any other psychotic disorder or organic mental disorder.
5. Has current suicidal ideation or homicidal ideation.
6. Has the need for maintenance or acute treatment with any psychoactive medication including anti-seizure medications and medications for ADHD.
7. Is currently taking medication known to affect alcohol intake (e.g., disulfiram, naltrexone, acamprosate, topiramate).
8. Has clinically significant medical problems such as cardiovascular, renal, GI, neurological (e.g. seizure disorder) or endocrine problems that would impair participation or limit medication ingestion.
9. Has past history of alcohol related medical illness such as gastrointestinal bleeding, pancreatitis, peptic ulcer, hepatic cirrhosis or alcoholic hepatitis.
10. Has hepatocellular disease indicated by elevations of SGPT (ALT) or SGOT (AST) greater than 2.5 times normal at screening.
11. Females of childbearing potential who are pregnant (by urine HCG), nursing, or who are not using a reliable form of birth control.
12. Has current charges pending for a violent crime (not including DUI related offenses).
13. Does not have a stable living situation.
14. Presence of ferrous metal in the body, as evidence by metal screening and self-report.
15. Severe claustrophobia or morbid obesity that preclude placement in the MRI scanner.
16. History of head injury with >2 minutes of unconsciousness.

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2016-03; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane Joseph, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Addiction Sciences Division-Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oxytocin/Alcohol Use Disorder | Placebo/Alcohol Use Disorder
Started | 5 | 6
Completed | 5 | 5
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxytocin/Alcohol Use Disorder | Placebo/Alcohol Use Disorder | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 25.2 [22 to 28] | 24 [22 to 27] | 24.6 [22 to 28]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 4 | 3 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 4 | 5 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Corticolimbic Functional Connectivity Based on fMRI Blood Oxygenation Level Dependent (BOLD) Response During the Stress Versus Neutral Conditions of the Montreal Imaging Stress Test Task Averaged Over the Second and Third Functional Runs
Description: Corticolimbic functional connectivity will be determined using psychophysiological interaction (PPI) modeling. The left and right amygdala will serve as seed regions. Connectivity of each seed region with the homologous orbitofrontal cortex region will be represented as a parameter estimate, yielding one parameter estimate for right amygdala-right orbitofrontal connectivity and one parameter estimate for left amygdala-left orbitofrontal connectivity per subject.
Time Frame: 60 minutes following medication (oxytocin or placebo)
Measure: Mean (Standard Deviation); unit: contrast of parameter estimates
Arm/Group | Oxytocin/Alcohol Use Disorder | Placebo/Alcohol Use Disorder
Number analyzed (Participants) | 5 | 5
contrast of parameter estimates
  Left amygdala left orbitofrontal connectivity | -.12723 (.103532) | -.04836 (.150718)
  Right amygdala right orbitofrontal connectivity | .042561 (.155865) | -.06624 (.240009)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Oxytocin/Alcohol Use Disorder | Placebo/Alcohol Use Disorder
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-04): https://cdn.clinicaltrials.gov/large-docs/33/NCT03610633/Prot_SAP_000.pdf